CLINICAL TRIAL: NCT00319878
Title: A Phase I/II Trial of Sirolimus (Rapamune) and Cyclosporine in Patients With Refractory Aplastic Anemia
Brief Title: Sirolimus and Cyclosporine for Treatment-Resistant Aplastic Anemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Office of Rare Diseases (ORD) (NIH)
Collaborators: Rare Diseases Clinical Research Network (Network)
Responsible Party: Ronald Paquette, MD, UCLA Division of Hematology/Oncology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDCRN 5403; U54RR019397-01 (NIH); BMF 5403
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Anemia, Aplastic
MeSH Terms: conditions — Anemia, Aplastic | interventions — Sirolimus; Cyclosporine

ARMS (1):
- 1 (Experimental): Participants will be treated with sirolimus and cyclosporine. In phase I, each dose cohort will initially enroll three patients. If no dose-limiting toxicity (DLT) is observed by Day 28 in any patient of a cohort, then 3 patients will be treated with the next highest sirolimus dose. If 1 out of 3 patients in any cohort experiences a DLT, then 3 more patients will be enrolled in that cohort. If no more patients have a DLT by Day 28, then sirolimus dose escalation will proceed. If one or more patients experience a DLT then that dose level will be considered to be the maximum tolerated sirolimus dose, and Phase II patients will be treated at the next lowest level. Cyclosporine will be given as a twice daily oral dose.
  Interventions: Drug: Sirolimus; Drug: Cyclosporine

INTERVENTIONS:
Drug: Sirolimus — Oral loading dose followed by a once daily dose:
  * Cohort 1: Loading Dose - 1.2 mg; Daily Dose - 0.4 mg
  * Cohort 2: % Dose Increase - 100%; Loading Dose - 2.4 mg; Daily Dose - 0.8 mg
  * Cohort 3: % Dose Increase - 67%; Loading Dose - 3.9 mg; Daily Dose - 1.3 mg
  * Cohort 4: % Dose Increase - 50%; Loading Dose - 6.0 mg; Daily Dose - 2.0 mg
Drug: Cyclosporine — Dose of 5 mg/kg divided as a twice daily oral dose

SUMMARY:
Aplastic anemia is a rare autoimmune disorder in which the bone marrow production of blood cells is greatly decreased or absent. Symptoms include fatigue, weakness, tiny reddish-purple marks on the skin, abnormal bruising, and bleeding from the gums, nose, or intestine. While some cases of aplastic anemia are caused by medications, toxic exposures, or inherited genes, most often the cause remains unknown. The purpose of this study is to determine the safety and efficacy of combining two drugs, sirolimus and cyclosporine, for treating individuals with aplastic anemia that has not responded to other treatments.

DETAILED DESCRIPTION:
The most successful treatment for aplastic anemia is bone marrow transplantation. However, few patients are eligible for this procedure. For others, treatment usually consists of immunosuppressive agents, such as antithymocyte globulin (ATG) and cyclosporine. Unfortunately, even with immunosuppressive therapy, relapse is common. New combinations of medications may offer alternative and more effective treatment options. Sirolimus and cyclosporine are two drugs routinely used to suppress the immune system and prevent rejection in patients who have received organ transplants. While cyclosporine has been proven effective for treating aplastic anemia, sirolimus has not been tested for this disease. This study will evaluate the safety and efficacy of sirolimus in combination with cyclosporine for treating individuals with aplastic anemia that has not responded to other treatments.

This study will last at least 6 months. Participants will first be screened to verify diagnosis of aplastic anemia. The screening will include a physical examination, blood test, bone marrow biopsy from the pelvic bone, and review of medications and medical history. Individuals who are eligible will then start the first treatment period. Participants will receive two medications: cyclosporine will be taken twice a day and sirolimus will be taken once a day. Depending on side effects, the doses of either drug may be temporarily stopped or lowered. On Day 1, blood will be drawn and females will undergo a pregnancy test. Subsequent study visits will occur weekly for the first month, every 2 weeks for 2 months, and then once a month for the remainder of the study. Each visit will include a physical examination, vital sign assessment, and review of side effects and medications. Blood tests will be performed weekly for the first 3 weeks, and then every 2 weeks.

After 6 months of treatment, if a participant has shown improvements in disease status without major side effects, the treatment will continue. Over time the doses may be lowered. If a participant has not improved while on the study medication, treatment will stop at 6 months. Whenever treatment is discontinued, the participant will again undergo a physical examination, blood tests, and bone marrow biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate or severe aplastic anemia with bone marrow cellularity of less than 25%
* Falls within one of the following descriptions at the time of the original diagnosis:

  1. For severe aplastic anemia, fulfills any two of the following three criteria: absolute neutrophil count less than 500/uL; absolute reticulocyte count less than 60,000/uL; and platelet count less than 20,000/uL
  2. For moderate aplastic anemia, fulfills any two of the following three criteria: absolute neutrophil count less than 1200/ul; hemoglobin less than 8 g/dL with corrected reticulocyte count less than 1%; and platelet count less than 60,000/uL (Note: Participants who have progressed from moderate to severe aplastic anemia prior to study entry will be classified as having severe aplastic anemia)
* Diagnosis of refractory aplastic anemia, as defined by a failure to achieve at least a partial response to ATG within 6 months of treatment. Individuals who had a prior response to ATG but who have relapsed and not responded to salvage ATG are eligible. Individuals with relapsed disease who are not candidates for salvage ATG because they experienced a serious or life-threatening complication prior to ATG are also eligible.
* A Karnofsky performance status of at least 60%
* Adequate organ function, as defined by creatine levels less than 1.5 times the upper limit normal (ULN), and liver function tests (AST, bilirubin) less than 2 times the ULN
* Women of childbearing age must be willing to use effective contraception throughout the study

Exclusion Criteria:

* Received ATG treatment less than 6 months prior to study entry
* Candidate for related allogeneic stem cell transplantation
* Active uncontrolled infection
* History of myelodysplastic syndrome or bone marrow cytogenetic abnormalities
* History of Fanconi's anemia or other congenital form of aplastic anemia
* Treatment with an investigational agent within 1 month of study entry
* HIV infection
* Pregnant or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-07 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of sirolimus and cyclosporine in each stratum of participants | Measured at Month 6

SECONDARY OUTCOMES:
Response rate | Measured at Months 3 and 6
Duration of hematologic response | Measured at Month 6
Rate of clonal disease evolution | Measured at Month 6
Survival | Measured at Month 6

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA Center for Health Sciences, Los Angeles, California
  - Lee Moffitt Cancer Center, Tampa, Florida
  - Taussig Cancer Center, Cleveland Clinic Foundation, Cleveland, Ohio
  - Penn State University Cancer Center, Hershey, Pennsylvania

REFERENCES:
- [Background] Maciejewski JP, Risitano AM. Aplastic anemia: management of adult patients. Hematology Am Soc Hematol Educ Program. 2005:110-7. doi: 10.1182/asheducation-2005.1.110. PMID 16304367
- [Background] Young NS. Immunosuppressive treatment of acquired aplastic anemia and immune-mediated bone marrow failure syndromes. Int J Hematol. 2002 Feb;75(2):129-40. doi: 10.1007/BF02982017. PMID 11939258
- [Background] Brodsky RA, Chen AR, Brodsky I, Jones RJ. High-dose cyclophosphamide as salvage therapy for severe aplastic anemia. Exp Hematol. 2004 May;32(5):435-40. doi: 10.1016/j.exphem.2004.02.002. PMID 15145211
- [Background] Paquette RL. Diagnosis and management of aplastic anemia and myelodysplastic syndrome. Oncology (Williston Park). 2002 Sep;16(9 Suppl 10):153-61. PMID 12380966